CLINICAL TRIAL: NCT05296226
Title: Effects of Dry Needling Versus Ischemic Compression on Pain, Range of Motion and Functional Disability in Chronic Neck Pain Patients With Trigger Points
Brief Title: Effects of Dry Needling Versus Ischemic Compression on Pain, Range of Motion and Finctional Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1085/2021
Record Dates: First submitted 2022-02-14; First posted 2022-03-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-02

CONDITIONS: Trigger Points
Keywords: dry needling; ischemic compression; trigger point; pain; range of motion; functional disability
MeSH Terms: conditions — Pain | interventions — Dry Needling; Acupressure; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling group (Experimental): dry needling is probably the most popular, trigger-point dry needling is an invasive procedure where a fine Needle or acupuncture needle is inserted into the skin and muscle Goniometry will be used to assess range ofmotion. Ischemic compression is one of the least invasive trigger point therapies.
  Interventions: Procedure: dry needling and ischemic compression
- ischemic compression group (Experimental): compression is one of the least invasive trigger point therapies. Ischemic compression is a mechanical treatment of myofascial trigger points that consists of application of sustained pressure for a long enough time to inactivate the trigger points. Pressure is sustained for 10 to 20 second
  Interventions: Procedure: dry needling and ischemic compression

INTERVENTIONS:
Procedure: dry needling and ischemic compression — dry needling is an invasive procedure where a fine Needle or acupuncture needle is inserted into the skin and muscle Ischemic compression is one of the least invasive trigger point therapies. Ischemic compression is a mechanical treatment of myofascial trigger points that consists of application of sustained pressure for a long enough time to inactivate the trigger points.
  Other Names: Exercises

SUMMARY:
Neck pain can occur from a number of conditions, most common is trigger points. Trigger points are of two point one is active and other is latent trigger point, hyperirritable spots located in a taut band of skeletal muscle. They produce pain locally and in a referred pattern and often accompany chronic musculoskeletal disorders. Acute trauma or repetitive micro trauma may lead to the development of stress on muscle fibers and the formation of trigger points Khadijeh Otadi and her colleague study in 2020, to compare immediate and short-term effects of combining dry needling patient education vs ischemic compression patient education for treating myofascial trigger points in office workers with neck pain. Both intervention groups had some positive immediate and short-term effects after 2 treatment sessions. However, Ischemic compression was more effective than Dry needling in the treatment of MTPs in office workers with neck pain.

Study design: randomized control trial (RCT) Settings: study will be conducted in DHQ hospital Okara physiotherapy department.

Duration of study: nine months after the approval of synopsis. Sample Size: 72 patients will be randomly divided into two equal groups of 36 each.

DETAILED DESCRIPTION:
A trigger points is composed of numerous so-called contraction knots. An individual contraction knot appears as a segment of a muscle fiber with extremely contracted sarcomeres and an increased diameter. 2 Trigger point can occur in a number of muscles but they are most common in rhomboid and trapezius muscles. The trapezius is a large paired trapezoid-shaped surface muscle that extends longitudinally from the occipital bone to the lower thoracic vertebrae of the spine and laterally to the spine of the scapula. The trapezius has three functional parts: upper, middle and inferiorfinding typically associated with a trigger point. 5 Active trigger point is any point that causes tenderness and referral pain pattern on palpation. Almost always central trigger points are active and some satellite trigger points are also active. Active trigger points usually produce referred pain and tenderness. In contrast, latent trigger points are foci of hyperirritability in a taut band of muscle, which are clinically associated with a local twitch response, tenderness and referred pain upon manual examination A researcher assessed in 2017, the immediate neurophysiological and clinical effects of DN in patients with upper trapezius MTrPs. The results of this study showed that one session of DN targeting active MTrPs appears to reduce hyperactivity of the sympathetic nervous system and irritability of the motor endplate. DN seems effective at improving symptoms and deactivating active MTrPs.

A study was conducted by Aleksandra k et al in 2018 that aimed to assess the effects of compression trigger point therapy on the stiffness of the trapezius muscle in professional basketball players. Study confirmed that a single treatment session of active myofascial trigger points with ischemic compression causes a decrease in muscle stiffness of the upper portion of the trapezius muscle. A decrease of muscle stiffness has been suggested to improve deficits in range of motion and thereby lower the risk of injuries among baseball players.

The patient's total session of treatment will be 4 weeks. The date will be collected by using questionnaire Neck disability index and Numerical pain rating scale. The number of patients will be randomly allocated 72 patients and 36 patients in each group. And they will be given session of dry needling and ischemic compression in 3 alternate days in a week. Results will be noted immediate after the treatment session then again note the response 3 days after treatment session and ultimately note the response 1 month after the treatment session

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-40 years.

  * Presence of palpable taut band in muscle.
  * Presence of a hypersensitive tender spot in the taut band.
  * Pain at least 8 points on a numeric pain scale (NPS)

Exclusion Criteria:

* History of fibromyalgia syndrome, whiplash injury, cervical spine surgery and fracture, cervical radiculopathy.
* Any systematic disease such as rheumatism, tuberculosis, cervical myelopathy, or multiple sclerosis.
* Peripheral nerve entrapment, fibromyalgia, hypermobility syndrome, shoulders diseases (tendonitis, bursitis, and capsulitis).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
NPRS | 4 weeks
  The number of patients will be 36. And they will be given session in 3 alternate days in a week. Results will be noted immediate after the treatment session then again note the response 3 days after treatment session and ultimately note the response 1 month after the treatment session. The patient's total session of treatment will be 4 weeks.
NDI | 4 weeks
  The number of patients will be 36. And they will be given session in 3 alternate days in a week. Results will be noted immediate after the treatment session then again note the response 3 days after treatment session and ultimately note the response 1 month after the treatment session. The patient's total session of treatment will be 4 weeks.
ROM | 4 weeks
  The number of patients will be 36. And they will be given session in 3 alternate days in a week. Results will be noted immediate after the treatment session then again note the response 3 days after treatment session and ultimately note the response 1 month after the treatment session. The patient's total session of treatment will be 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: RABIA ASHIQ, PT, Principal Investigator — University of Lahore
Locations (1):
- Hafiz Ijaz Bhaati, Okara, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided